CLINICAL TRIAL: NCT02088645
Title: 177Lu-PP-F11N for Receptor Targeted Therapy and Imaging (Theranostics) of Metastatic Medullary Thyroid Cancer - a Pilot and a Phase I Study.
Brief Title: 177Lu-PP-F11N for Receptor Targeted Therapy and Imaging of Metastatic Thyroid Cancer.
Acronym: Lumed
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Krebsforschung Schweiz, Bern, Switzerland (Other); Center for Proton Therapy, Paul Scherrer Institute, Villigen,Switzerland (Other); University Hospital, Zürich (Other); University Hospital Freiburg (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KFS-3170-02-2013
Record Dates: First submitted 2014-02-19; First posted 2014-03-17 (Estimated); Last update posted 2025-02-24 (Actual); Status verified 2024-12

CONDITIONS: Thyroid Cancer, Medullary; Neuroendocrine Tumor of the Lung Grade 1 and 2; Neuroendocrine Tumor of the Thymus Grade 1 and 2; Neuroendocrine Tumor GEP Grade 1-3
Keywords: Calcitonin; Medullary thyroid carcinoma; Peptide receptor radionuclide therapy; Gastrin; Cholecystokinin-2 receptor; Neuroendocrine tumor
MeSH Terms: conditions — Thyroid cancer, medullary; Carcinoma, Medullary; Neuroendocrine Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Phase 0: One arm; Phase I: One arm (Experimental): Phase 0: 6 patients, intravenous application of 2 x 1 gigabequerel (GBq) 177Lu-PP-F11N with and without Physiogel (crossover)
  Phase I: expected 12 - 18 patients, intravenous application of max. 6 x 7-8 GBq 177Lu-PP-F11N (increasing number of applications by one in groups of three patients). All patients with or without Physiogel, depending on the results of the phase 0 study.
  Interventions: Drug: 177Lu-PP-F11N

INTERVENTIONS:
Drug: 177Lu-PP-F11N
  Other Names: Minigastrin analogue; Gastrin analogue; Cholecystokinin-2 receptor ligand

SUMMARY:
The purpose of this study is to determine the use of 177Lu-PP-F11N for imaging and therapy of patients with advanced medullary thyroid carcinoma (MTC). 177Lu-PP-F11N is a gastrin analogon, binding to cholecystokinin-2 receptors. This receptors show an overexpression on more than 90 % of medullary thyroid carcinomas.

In the pilot (phase 0) study investigators will correlate the tumour detection rate with the surgery and histology (proof of concept study). Furthermore, kidney protection and dosimetry studies will be performed in order to determine the kidney protection protocol and starting activity for the dose escalation study in the following, dose escalation (phase I) study. In the phase I study investigators will determinate the maximum tolerated dose of 177Lu-PP-F11N in patients with MTC. Furthermore, correlation with tumour radiation dose and treatment response as well as organ radiation doses and maximal tolerated dose will be performed in order to allow prospective individual patient tailored therapy planning. In the phase I study, participation is additionally possible for patients with well differentiated GEP-NET (grade 1-3) with a Ki67 index of up to 55% or NET of the lung or thymus (grade 1 and 2).

ELIGIBILITY:
Inclusion Criteria:

Phase 0 study

* Advanced MTC with elevated levels of calcitonin (> 100 pg/ml) and/or calcitonin-doubling time < 24 months before or after total thyroidectomy or
* Patients with well differentiated GEP-NET (grade 1-3) with a Ki67 index of up to 55% or NET of the lung or thymus (grade 1 and 2) with low or missing expression of SST2-receptor and progressive disease within the last 6 months according to RECIST 1.1
* Age > 18 years
* Informed consent

Phase I study

* Diagnostic, contrast medium enhanced CT scan neck/thorax/abdomen, not older than 4 weeks
* Advanced MTC with elevated levels of calcitonin (> 100 pg/ml) and/or calcitonin-doubling time < 24 months before or after total thyroidectomy- Age > 18 Years
* Informed consent
* Curative surgical therapy not possible

Exclusion Criteria:

Phase 0 study

* Medication with Vandetanib 3 weeks before the study and during the study
* Renal failure (calculated glomerular filtration rate (GFR) < 60 ml/min per 1.73 m2 body surface).
* Bone marrow failure (thrombocytes < 70 000/μl, leucocytes < 2 500/μl, hemoglobin < 8 g/dl).
* Pregnancy and breast feeding
* Knows allergic reaction on Physiogel or other gelatine products
* Known, serious side reaction in the case of a former application of pentagastrin
* Active, second malignancy oder remission after second malignancy < 5 years

Phase I study

* Medication with Vandetanib 3 weeks before the study and during the study
* Renal failure (calculated GFR < 50 ml/min per 1.73 m2 body surface).
* Bone marrow failure (thrombocytes < 100 000/μl, leucocytes < 3 000/μl, hemoglobin < 10 g/dl).
* Pregnancy and breast feeding
* Known, serious side reaction in the case of a former application of pentagastrin
* Active, second malignancy oder remission after second malignancy < 5 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2015-04; Primary Completion 2026-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Phase 0: Scintigraphic visualisation rate | up to 4 weeks
  Phase 0 study: Evaluation of the scintigraphic visualisation of metastases after test injection, verification of 177Lu-PP-F11N uptake in metastases and correlation with surgery/histology if possible (poof of principle study).
Phase I: Maximum tolerated dose | Up to 9 months
  Phase I study: Determination of the maximum tolerated dose (MTD)

SECONDARY OUTCOMES:
Phase 0: Tumour-to-kidney radiation doses | 8 and 16 weeks
  Evaluation of the kidney radiation dose and the tumour-to-kidney radiation dose ratios with and without kidney protection (Physiogel). Composite measure.
Phase 0: Radiation doses | 8 and 16 weeks
  Calculation of tumour and organ radiation doses.
Phase 0: In vivo stability | 8 and 16 weeks
  Evaluation of in vivo stability of 177Lu-PP-F11N.
Phase 0: Metabolites | 8 and 16 weeks
  Measurement of the metabolites of 177Lu-PP-F11N with and without Physiogel infusion.
Phase I: Side reactions | 8, 16 and 24 weeks
  Evaluation of side reactions of 177Lu-PP-F11N.
Phase 1: Biochemical response | For the duration of 24 months.
  Evaluation of biochemical response (decrease of calcitonin and calculation of calcitonin doubling time).
Phase I: Morphological response | 0, 3 and 12 months
  Evaluation of morphological therapy response (RECIST criteria).
Phase I: Tumour detection rate | 8, 16 and 24 weeks
  Determination of the tumour detection rate and correlation with surgery/histology, if possible.
Phase I: Organ radiation doses | 8, 16 and 24 weeks
  Calculation of organ radiation doses after therapy and correlation with the determined MTD (composite measure).
Phase 1: Overall survival | Up to 5 years
  Determination of overall survival of patients after therapy.
Phase 1: In vivo stability | 8, 16 und 24 weeks
  Evaluation of in vivo stability of 177Lu-PP-F11N.
Phase 1: Metabolites | 8, 16 and 24 weeks
  Measurement of the metabolites of 177Lu-PP-F11N.

CONTACTS AND LOCATIONS:
Overall Officials: Christof Rottenburger, Dr. med., Principal Investigator — University Hospital, Basel, Switzerland; Damian Wild, Prof Dr Dr, Study Director — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Clinic for radiology and nuclear medicine, Basel, Switzerland

REFERENCES:
- [Background] Sauter AW, Mansi R, Hassiepen U, Muller L, Panigada T, Wiehr S, Wild AM, Geistlich S, Behe M, Rottenburger C, Wild D, Fani M. Targeting of the Cholecystokinin-2 Receptor with the Minigastrin Analog 177Lu-DOTA-PP-F11N: Does the Use of Protease Inhibitors Further Improve In Vivo Distribution? J Nucl Med. 2019 Mar;60(3):393-399. doi: 10.2967/jnumed.118.207845. Epub 2018 Jul 12. PMID 30002107
- [Background] Rottenburger C, Nicolas GP, McDougall L, Kaul F, Cachovan M, Vija AH, Schibli R, Geistlich S, Schumann A, Rau T, Glatz K, Behe M, Christ ER, Wild D. Cholecystokinin 2 Receptor Agonist 177Lu-PP-F11N for Radionuclide Therapy of Medullary Thyroid Carcinoma: Results of the Lumed Phase 0a Study. J Nucl Med. 2020 Apr;61(4):520-526. doi: 10.2967/jnumed.119.233031. Epub 2019 Sep 13. PMID 31519804
- See also: Homepage University Hospital Basel — https://www.unispital-basel.ch/en